CLINICAL TRIAL: NCT05555706
Title: A Phase II/III Study to Evaluate the Efficacy and Safety of B013 in Combination With Nab-Paclitaxel in First-line Treatment for Patients With Previously Untreated Locally Advanced or Metastatic Triple Negative Breast Cancer
Brief Title: Study of B013 and Nab-Paclitaxel for Locally Advanced or Metastatic Triple Negative Breast Cancer
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Shanghai Jiaolian Drug Research and Development Co., Ltd (Industry)
Collaborators: Shanghai Pharmaceuticals Holding Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B013-301
Record Dates: First submitted 2022-09-22; First posted 2022-09-27 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-01

CONDITIONS: Triple Negative Breast Cancer (TNBC)
MeSH Terms: conditions — Triple Negative Breast Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- B013+ Nab-Paclitaxel (Experimental): B013 at a fixed dose of 600 milligrams via intravenous (IV) infusion on Days 1 and 15 of the first 28-day cycle, then on Day 1 of each subsequent 28-day cycle.
  Nab-Paclitaxel 100 mg/m^2 is administered weekly on Days 1, 8, 15 of each 28-day cycle.
  Interventions: Drug: B013+Nab-Paclitaxel

INTERVENTIONS:
Drug: B013+Nab-Paclitaxel — B013 at a fixed dose of 600 milligrams via intravenous (IV) infusion on Days 1 and 15 of the first 28-day cycle, then on Day 1 of each subsequent 28-day cycle.
  Nab-Paclitaxel 100 mg/m^2 is administered weekly on Days 1, 8, 15 of each 28-day cycle.

SUMMARY:
This Phase II/III study assessed the efficacy, safety, pharmacokinetics, and immunogenicity of B013 administered with nab-paclitaxel in participants with locally advanced or metastatic triple negative breast cancer (TNBC) who have not received prior systemic therapy for metastatic breast cancer (mBC).

ELIGIBILITY:
Inclusion Criteria:

1. Women or men aged 18 -75 years
2. Locally advanced or metastatic triple negative breast cancer (TNBC)
3. No prior chemotherapy or targeted systemic therapy for inoperable locally advanced or metastatic TNBC
4. ECOG performance status of 0 or 1
5. Patient must have measurable or evaluable disease as defined by RECIST v1.1. Measurable lesions will be confirmed by radiographic imaging (CT or MRI)

Exclusion Criteria:

1. Previous treatment is eligible.
2. Spinal cord compression not definitively treated with surgery and/or radiation prior to study entry
3. Known central nervous system (CNS) disease
4. Uncontrolled pleural effusion, pericardial effusion, or ascites Patients
5. Uncontrolled tumor-related pain prior to study entry
6. The patient has a history of another malignancy within 5 years prior to study entry, except adequately treated non-melanotic skin cancer, carcinoma in situ of the cervix or Papillary carcinoma of the thyroid
7. Pregnancy or lactation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2022-12-06 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Objective response rate (ORR)(phase Ⅱ) | Baseline up to approximately 18 months
  tumor response will be evaluated according to the Response Evaluation Criteria Solid Tumors (RECIST) criteria version 1.1.
Progression-free survival (PFS)(IRC) (phase Ⅲ) | Baseline up to approximately 18 months
  from the start date of study treatment to the date of progression disease or death , whichever occurred first.

SECONDARY OUTCOMES:
Disease control rate (DCR) | 18 months
  DCR was defined as the percentage of patients who have achieved complete response, partial response and stable disease
Duration of remission (DOR) | 18 months
  DOR was defined for participants who had an objective response as the time from the first occurrence of a documented unconfirmed response (CR or PR) to the date of disease progression per RECIST v1.1 or death from any cause
Time to Response (TTR) | 18 months
  Defined as the interval from the start of study therapy to the first documentation of an objective response
Overall Survival (OS) | 3years
  Determination of the overall survival times of all patients
Drug concentration in plasma | 18 months
  Determination of drug concentration in plasma of all patients
Incidence of Treatment-Emergent Adverse Events | 3years
  Adverse event type, incidence, duration, correlation with study drug

CONTACTS AND LOCATIONS:
Overall Officials: Shusen Wang, Principal Investigator — Affiliated Cancer Hospital, Sun Yat-sen University; Huiping Li, Principal Investigator — Peking University Cancer Hospital & Institute
Locations (13):
- China (13):
  - Affiliated Cancer Hospital, Sun Yat-sen University, Guangzhou, Guangdong
  - Guangxi Medical University Cancer Hospital, Nanning, Guangxi
  - Hainan cancer Hospital, Haikou, Hainan
  - The First Affiliated Hospital of henan University of Science and Technoloy, Luoyang, Henan
  - Xiangyang Central Hospital, Xiangyang, Hubei
  - The Central Hospital of Yongzhou, Yongzhou, Hunan
  - Huai'an First People's Hospital, Huai'an, Jiangsu
  - Sichuan Cancer Hospital, Chengdu, Sichuan
  - The second people's hospital of neijiang, Neijiang, Sichuan
  - Yunnan Cancer Hospital, Kunming, Yunnan
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang
  - Peking University Cancer Hospital, Beijing
  - Tianjin medical university cancer institute&hospital, Tianjin